CLINICAL TRIAL: NCT02869880
Title: Trial of Enhanced Pre-Consent Discussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); ImproveCareNow (ICN) (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Ellen A. Lipstein MD, MPH, Assistant Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015-9033
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Pediatric Crohn's Disease
MeSH Terms: conditions — Pediatric Crohn's disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Pre-consent Discussion (Active Comparator): Standard pre-consent discussion for a clinical trial.
  Interventions: Other: Standard Pre-consent Discussion
- Enhanced Pre-consent Discussion (Experimental): The enhanced pre-consent discussion intervention is a tool that includes both textual and graphical information regarding the trial and an interactive component designed to initiate and facilitate conversations between all parties in the decision-parent, patient, healthcare provider and research staff.
  Interventions: Other: Enhanced Pre-Consent Discussion

INTERVENTIONS:
Other: Enhanced Pre-Consent Discussion — The enhanced pre-consent discussion intervention is a tool that includes both textual and graphical information regarding the trial and an interactive component designed to initiate and facilitate conversations between all parties in the decision-parent, patient, healthcare provider and research staff.
  Arms: Enhanced Pre-consent Discussion
Other: Standard Pre-consent Discussion — Standard pre-consent discussion for a clinical trial
  Arms: Standard Pre-consent Discussion

SUMMARY:
Nested within the COMBINE pragmatic clinical trial, the investigators will conduct a cluster randomized controlled trial to determine whether, in parents (of children with Crohn's Disease) or patients > 18 years old being approached for trial participation, a pre-consent discussion enhanced with decision aids is more effective than the standard pre-consent discussion in transferring knowledge to parents/patients related to trial participation.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child who is eligible for the COMBINE trial (ClinicalTrials.gov Identifier: NCT02772965)
* Patient who is eligible for the COMBINE trial (ClinicalTrials.gov Identifier: NCT02772965)

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Knowledge Related to Trial Participation | prior to consent
  Number correct on 5-item Knowledge Related to Trial Participation survey

SECONDARY OUTCOMES:
Rate of enrollment | at consent
Support subscale of decision conflict scale | prior to consent

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Lipstein, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No